CLINICAL TRIAL: NCT05074264
Title: Optimization of Screening Algorithms for Cervical and Anal High-Grade Squamous Intraepithelial Lesions in People Living With HIV in Mexico and Puerto Rico
Brief Title: Screening Algorithms for Cervical and Anal High-Grade Squamous Intraepithelial Lesions in People With HIV in Mexico and Puerto Rico
Acronym: CAMPO-101
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); US-Latin American-Caribbean HIV/HPV-Cancer Prevention Clinical Trials Network (ULACNet) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21622; NCI-2020-13805 (Registry Identifier: NCI Clinical Trial Reporting Program (CTRP)); ULACNet-101 (Other: Division of Cancer Prevention); U54CA242646 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: AIDS-Related Anal Carcinoma; AIDS-Related Cervical Carcinoma; High Grade Anal Intraepithelial Neoplasia; High Grade Cervical Intraepithelial Neoplasia; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Biopsy; Colposcopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Imaging, biospecimen collection, anoscopy and/or colposcopy (Experimental): Patients undergo collection of cervical images (if applicable), 3 cervical anal swabs (if applicable) and 3 anal swabs for real-time testing of HPV or hrHPV over 90 minutes. Patients with a positive HPV or hrHPV test on undergo biopsies of visible lesions. Patients with a negative hrHPV test on their cervical swab may undergo a colposcopy. Patients with a positive hrHPV test on their anal swab undergo high-resolution anoscopy at a later visit within 1 month. Patients with a negative hrHPV on their anal swabs may undergo a high-resolution anoscopy and biopsies of visible lesions, and those with a positive anal cytology for LSIL or worse undergo a high-resolution anoscopy and biopsies within 1 month. Patients may be given a diagnosis and treatment at the second visit. Patients diagnosed with HSIL may undergo SOC treatment or enroll in additional studies when they are open to accrual
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection - Anal; Procedure: Biospecimen Collection - Cervical; Procedure: Colposcopy; Procedure: High Resolution Anoscopy; Procedure: Imaging Technique

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
Procedure: Biospecimen Collection - Anal — Undergo collection of anal swabs
  Other Names: Biological Sample Collection; Biospecimen Collection
Procedure: Biospecimen Collection - Cervical — Undergo collection of cervical swabs
  Other Names: Biological Sample Collection; Biospecimen Collection
Procedure: Colposcopy — Undergo colposcopy
Procedure: High Resolution Anoscopy — Undergo high-resolution anoscopy
  Other Names: HRA
Procedure: Imaging Technique — Undergo cervical imaging
  Other Names: Diagnostic Imaging Technique; Imaging; Imaging Procedures; Medical Imaging

SUMMARY:
This clinical trial aims to find what different tests work best to find high-grade squamous intraepithelial lesions (HSIL) in the cervix or anus in patients living with human immunodeficiency virus (HIV). Patients with HIV are at high risk of becoming infected with human papillomavirus (HPV) in the cervix or anus where it can turn into cancer over several years. HPV causes changes to the cervix and anus, known as HSIL. This means that there is an area of abnormal tissue on the top layers of the cervix or anus. It is considered cervical or anal cancer if the abnormality spreads down into the layers of tissue below the top. If found early, many cases of HSIL can be treated before turning into cancer. Screening for cervical or anal cancer detection or HSIL associated with HPV may result in earlier treatment, if necessary, for patients living with HIV.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the most efficient algorithm combining point-of-care (POC) HPV-based screening with several triage alternatives: cytology, E6 and/or E7 oncoprotein detection and S5 methylation, to improve the current screening program for detection of anogenital HPV-related cancers and pre-cancers, in men and women living with HIV in Mexico and Puerto Rico.

EXPLORATORY OBJECTIVE:

I. Evaluate artificial intelligence-based algorithms based on cell-phone images of the cervix for their sensitivity, specificity, and negative and positive predictive values for cervical cancers and precancers in women living with HIV in Mexico and Puerto Rico.

II. Evaluate the HPV agreement/concordance between cervicovaginal samples collected by participants and cervical samples collected by clinicians.

OUTLINE: Patients receive standard medical procedures based on anatomy at time of enrollment.

GROUP I (WOMEN LIVING WITH HIV (WLWH)): Patients undergo collection of cervical images, 3 cervical anal swabs and 3 anal swabs for real-time testing of high-risk (hr) HPV over 90 minutes. Patients with a positive hrHPV test on their cervical swab undergo colposcopy and biopsies of visible lesions. Patients with a negative hrHPV test on their cervical swab may undergo a colposcopy. Patients with a positive hrHPV test on their anal swab undergo high-resolution anoscopy at a later visit within 1 month. Patients with a negative hrHPV on their anal swabs may undergo a high-resolution anoscopy and biopsies of visible lesions, and those with a positive anal cytology for low-grade squamous intraepithelial lesion (LSIL) or worse undergo a high-resolution anoscopy and biopsies within 1 month. Patients may be given a diagnosis and treatment at the second visit. Patients diagnosed with HSIL may undergo standard of care (SOC) treatment or enroll in additional studies when they are open to accrual.

GROUP II (MEN LIVING WITH HIV (MLWH)): Patients undergo collection of 3 anal swabs for real-time testing of high-risk HPV over 90 minutes. Patients with a positive hrHPV test undergo high-resolution anoscopy with biopsies of visible lesions. Patients with hrHPV negative test may undergo high-resolution anoscopy. Patients may be given a diagnosis and treatment at the second visit. Patients diagnosed with HSIL may undergo SOC treatment or enroll in additional studies when they are open to accrual.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care provider
  * Documentation of receipt of antiretroviral therapy (ART) by a licensed health care provider (Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name. Receipt of at least two agents is required; each component agent of a multi-class combination ART regimen will be counted toward the 2-agent requirement, excepting receipt of a pre-exposure prophylaxis (PrEP) regimen alone [e.g., Truvada], which is exclusionary);
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating > 1000 RNA copies/mL
  * Any locally licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay
  * NOTE: A "licensed" assay refers to a United States (U.S.) Food and Drug Administration (FDA)-approved assay or an assay approved by the relevant local health authority
* Age 21 years or older. Cervical HSIL/cancer screening does not usually begin until 20 years of age or older. Also, anal HSIL/cancer screening among high risk individuals such as people living with HIV is recommended for those 25 years of age or older. Children under the age of 18 are at low risk of developing cervical or anal HSIL/cancer and will not benefit from the kind of screening planned for this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky score >= 70%)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have undergone hysterectomy
* History of anal cancer, penile, vulvar, vaginal, or cervical cancer
* Potential participants who received prior treatment of anal, cervical, penile, vaginal, or vulvar lesions within 18 months of study enrollment
* Inability in the opinion of the study investigator of the participant to comply with study requirements
* Participants who are pregnant (a urine pregnancy test will be provided to participants aged 60 years or less) or within 2 months being post-partum

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1586 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Most efficient algorithm for detection of anogenital human papillomavirus (HPV)-related cancers and high-grade squamous intraepithelial lesions (HSIL) | Up to 3 years
  Will assess a screening algorithm with an optimal combination of: point of care high-risk (hr) HPV testing, extended hrHPV genotyping, cytology, progression markers protein E6 and S5 methylation score, to identify cervical and/or anal HSIL or cancer. Different contingency tables will be prepared to describe the statistical relationship between hrHPV infection and HSIL positive status. Using the Bayes Rule, the predicted values will the computed using the prevalence of HSIL positive (overall and per country), where prevalence is the probability of currently being HSIL positive regardless of the duration of time one has the disease. The positive Diagnostic Likelihood Ratios (DLR) and the Negative Diagnostic Likelihood Ratio will be computed to determine the best strategy combining sensitivity and specificity. The 95% confidence intervals of DLR+ will be computed using the log approach.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- Mexico (3):
  - Condesa Specialized Clinic, Mexico City, Mexico City
  - Condesa Iztapalapa Specialized Clinic, Mexico City, Mexico City
  - Instituto Nacional de Cancerologia (INCan), Mexico City, Mexico City
- University of Puerto Rico Comprehensive Cancer Center, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No